CLINICAL TRIAL: NCT06706752
Title: A Randomized, Blinded, Placebo-controlled Trial of Shengbai Oral Formula to Assess Safety and Alleviation of Adverse Effects in Patients With Cancer Undergoing Chemotherapy
Brief Title: A Study of Shengbai Oral Formula to Assess Safety and Alleviation of Adverse Effects in Cancer Patients Undergoing Chemotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sutter Health (Other)
Responsible Party: Principal Investigator, Amy Matecki, Principal Investigator and Holistic/Integrative Medicine Physician, Sutter Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2052995
Record Dates: First submitted 2024-11-21; First posted 2024-11-27 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group (Experimental)
  Interventions: Dietary Supplement: Shengbai Oral Formula
- Placebo Group (Placebo Comparator)
  Interventions: Other: Inactive Placebo

INTERVENTIONS:
Dietary Supplement: Shengbai Oral Formula — Shengbai Oral Formula contains 11 herbs: Folium Epimedii, Fructus Lycii, Radix Astragali, Caulis Spatholobi, Radix Rubiae, Rhizoma Phragmitis, Fructus Psoraleae, Radix Angelicae Sinensis, Radix Ophiopogonis,, Radix et Rhizoma Glycyrrhizae, Radix Aconiti Lateralis Preparata (Processed). It is taken by mouth three times per day for 14 days.
  Arms: Treatment Group
Other: Inactive Placebo — Inactive placebo will be taken by mouth three times per day for 14 days.
  Arms: Placebo Group

SUMMARY:
The goal of this clinical trial is to assess whether Shengbai Oral Formula is a viable option for treatment of fatigue, pain, and neutropenia in patients undergoing their third cycle of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years of age
2. A cancer diagnosis and scheduled to undergo at least three rounds of chemotherapy for curative or palliative intent
3. Chemotherapy is given at a minimum of every 2 weeks
4. At least 30 days past radiation therapy
5. Nonpregnant and use of method of contraception per the treating clinician standard of care
6. Life expectancy > 3 months
7. Stable on all herbal or complementary therapeutics for the past 30 days and agree to not include new complementary therapeutics until after study completion
8. Baseline ECOG ≤ 2
9. In the opinion of the investigator, the subject will be compliant and have a high probability of completing the study including all scheduled evaluations and required tests

Exclusion Criteria:

1. Abnormal ALT/AST: > 2.5 to 3 times normal range
2. eGFR <60
3. Platelets < 75,000
4. Hb <8.0
5. ANC <1000
6. Documentation of a bone marrow transplant
7. Documentation of brain metastases, diagnosis with other cancer, except skin cancer history with basal cell carcinoma, squamous carcinoma
8. Documentation of current seizure disorder
9. Documentation of new cardiac arrhythmias and myocardial infarction
10. Any active bacterial or viral infection, pneumonia, sepsis, active gastric ulcer, gastritis, nonhealing wound, intractable nausea or vomiting, diarrhea, bleeding disorder
11. Hyperthyroidism, connective tissue disease including systemic lupus erythematous, rheumatoid arthritis
12. Documentation of a current drug abuse disorder
13. Current participation in other clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Brief Fatigue Inventory | 14 days
  The Brief Fatigue Inventory (BFI) is used to assess the severity and impact of fatigue, including cancer-related fatigue. Fatigue scores on the BFI are categorized as Mild (1-3), Moderate (4-6), and Severe (7-10).

CONTACTS AND LOCATIONS:
Locations (1):
- Sutter Health, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No